CLINICAL TRIAL: NCT03645070
Title: A Prospective Randomized Study on the Effect of Oesophageal Temperature Monitoring on the Incidence of Esophageal Lesions After Left Atrial Ablation for the Treatment of Atrial Fibrillation.
Brief Title: Randomized Study on the Effect of Oesophageal Temperature on the Incidence of Esophageal Lesions After AF Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Circa Scientific, Inc. (Industry)
Responsible Party: Principal Investigator, Mauricio Ibrahim Scanavacca, Arrhythmia Clinical Unit Director, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Arrit-Incor-2
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Arrhythmias; Atrial Fibrillation; Esophageal Ulcer
Keywords: atrial-esophageal fistula; radiofrequency ablation; Atrial Fibrillation ablation
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- No probe (No Intervention): Twenty patients will be allocated to this group, which will have no esophageal temperature monitoring technique
- Single probe thermometer (Active Comparator): Twenty patients will be allocated in this group, in which there will be monitoring of esophageal temperature during radiofrequency applications in the posterior wall of the left atrium, with unipolar thermometer.
  Interventions: Device: Single probe thermometer
- Multi-probe (Active Comparator): Twenty patients will be allocated in this group, in which there will be esophageal temperature monitoring during radiofrequency applications in the posterior wall of the left atrium, with a multipolar and self expandable thermometer.
  Interventions: Device: multipolar and self expandable thermometer

INTERVENTIONS:
Device: multipolar and self expandable thermometer — Will be evaluated if a multipolar and self expandable thermometer is superior to no probe or to single probe thermometer at prevention of esophageal thermal injury.
  Other Names: CIRCA's S-CATH™ Esophageal Temperature Monitoring System
  Arms: Multi-probe
Device: Single probe thermometer — Will be evaluated if a single probe thermometer is superior to a multipolar and self expandable thermometer or to no probe thermometer at prevention of esophageal thermal injury
  Arms: Single probe thermometer

SUMMARY:
It's a randomized pilot study to evaluate the incidence of esophageal thermal injury after left atrial ablation for the treatment of atrial fibrillation according to three different strategies of esophageal temperature monitoring.

These patients will be divided into 3 groups with different strategies of esophageal temperature monitoring: group 1 without monitoring, group 2 monitoring with single probe thermometer and group 3 monitoring with multi-probe thermometer.

The primary end point will be the incidence of esophageal lesions assessed by upper endoscopy.

DETAILED DESCRIPTION:
This is a randomized pilot study on the effect of oesophageal temperature monitoring on the esophageal thermal injury after left atrial ablation for the treatment of atrial fibrillation (AF).

Sixty patients with paroxysmal AF or persistent and without previous AF ablation with indication of AF ablation will be selected to be included at the study.

After informed consent, these patients will be randomized in 3 groups with different strategies of esophageal protection for radiofrequency application in the posterior wall of the left atrium, by randomization in a ratio of 1: 1: 1 between groups.

Group I: no esophageal temperature monitoring technique. Group II: monitoring of esophageal temperature during radiofrequency applications in the posterior wall of the left atrium, with unipolar thermometer.

Group III: oesophageal temperature monitoring during radiofrequency applications in the posterior wall of the left atrium, with a multipolar and self expandable thermometer.

The primary end point will be the incidence of esophageal lesions assessed by upper endoscopy that will be done in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal or persistent AF, diagnosed by electrocardiogram, 24-hour Holter, or monitors of implantable or non-implantable events, with at least one episode of AF up to 12 months before the procedure. Patients should be willing and able to sign an informed consent form, and to undergo all procedures described in both the study protocol and the consent form.

Exclusion Criteria:

* Atrial thrombus in the left atrium, history of AF ablation, history of cardiac surgery, contraindication to anticoagulation, permanent AF, New York Heart Association functional class III or IV, stroke in the last 3 months, pregnancy, history blood clotting abnormalities, previous oesophageal surgery, or advanced chronic kidney disease (creatinine > 2.5 mg/dl).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Incidence of esophageal lesions | Within three days after the ablation procedure.
  Incidence of esophageal lesions evaluated by upper digestive endoscopy

SECONDARY OUTCOMES:
Rate of recurrence of AF | Six months
  Rate of recurrence of AF after ablation assessed by ECG, Holter 24 hours or clinically.
Isolation rate of pulmonary veins at the end of ablation. | End of the procedure
  Will be assessed the rate of pulmonary veins isolation
Duration of the AF ablation procedure | End of the procedure
  Will be assessed the duration of the AF ablation that will start at the time of the first radio-frequency lesion until the last one.
Incidence of atrio-esophageal fistulas | Six months
  Incidence of atrio-esophageal fistulas after AF ablation
Difference in the size of the esophageal lesions | Within three days
  Difference in the size of the esophageal lesions evaluated in the upper digestive endoscopy according to the different groups
Persistence of esophageal lesions in the second upper endoscopy. | Between 3 to 30 days of the procedure
  If necessary, the patients with esophageal lesions will be submitted to another upper endoscopy, and the persistence of esophageal lesions will be assessed
Maximum esophageal temperature reached during ablation. | During procedure.
  In the groups with esophageal temperature monitoring, the maximum esophageal temperature will be assessed and evaluated between two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio I Scanavacca, MD, PhD, Principal Investigator — Instituto do coração - HC/FMUSP
Locations (1):
- Arrhythmia Clinical Unit - Instituto do Coração - HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moura DMC, Pereira RAR, Pisani CF, Wu TC, Chokr MO, Hardy CA, Melo SL, Darrieux FCDC, Hachul DT, Scanavacca MI. Esophageal Temperature Monitoring during Atrial Fibrillation Ablation: A Randomized Study. Arq Bras Cardiol. 2025 Jun;122(7):e20250056. doi: 10.36660/abc.20250056. English, Portuguese. PMID 40767688